CLINICAL TRIAL: NCT00670956
Title: Investigation of Prenatal Steroids for Treatment of Prenatally Diagnosed CCAMs
Brief Title: Prenatal Steroids for Treatment of Congenital Cystic Adenomatoid Malformations (CCAM)
Acronym: CCAM Steroids
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Recruitment has been poor. Study drug is being offered as part of standard care of women carrying a pregnancy diagnosed with CCAM
Sponsor: University of California, San Francisco (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other); Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 10-03705
Record Dates: First submitted 2008-04-30; First posted 2008-05-02 (Estimated); Results first posted 2015-03-30 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Congenital Cystic Adenomatoid Malformation
Keywords: prenatal steroids; hydrops; congenital cystic adenomatoid malformation of the lung; prenatal intervention; betamethasone; prenatal diagnosis
MeSH Terms: conditions — Cystic Adenomatoid Malformation of Lung, Congenital; Edema | interventions — Betamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Study Group (Active Comparator): STEROID: Betamethasone; 12 mg intramuscularly x 2 doses 24 hours apart
  Interventions: Drug: Betamethasone
- Placebo Group (Placebo Comparator): PLACEBO: IM x 2 doses 24 hours apart
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Betamethasone — 12 mg intramuscularly x 2 doses 24 hours apart
  Arms: Active Study Group
Drug: Placebo — PLACEBO: IM x 2 doses 24 hours apart
  Arms: Placebo Group

SUMMARY:
Congenital cystic adenomatoid malformations (CCAMs) are theorized to be growing immature lung tissue. Administration of maternal steroids in the mid-trimester may stop the growth or decrease the size of the CCAM, thus increasing normal lung tissue and improving survival in fetuses with large CCAMs. This is a prospective, blinded, randomized trial comparing administration of a single course of antenatal steroids (Betamethasone) to control (i.e., placebo). The primary outcome variable will be incidence of hydrops. One month postnatal survival and relative size of the CCAM as determined by CCAM volume:head circumference ratio (CVR) between treatment/no treatment groups will be secondary outcome variables. Change in size of CCAM will be serially followed for both groups with individual growth curves being plotted prenatally and these will be compared with pathology weigh and volume to evaluate treatment effect. Other prenatal data collected will include: incidence of polyhydramnios, incidence of premature rupture of membranes, incidence of material complications. We will also compare mode of delivery, postnatal respiratory compromise, need for resection in the first week of life, and occurrence of complications during newborn administration

ELIGIBILITY:
Inclusion Criteria:

* GA < 26 weeks
* Maternal age > 18 years of age
* Singleton pregnancy
* Normal chromosomes
* CCAM volume to head circumference ratio (CVR) > 1.4
* No maternal medical/surgical contraindications
* No evidence of hydrops
* Not previously randomization

Exclusion Criteria:

* Maternal diabetes or use of insulin
* Preterm labor
* Multiple congenital anomalies with CCAM
* Chromosomal anomaly with CCAM
* Multiple gestation pregnancy with CCAM
* Not willing to be randomized
* Unable or unwilling to return to UCSF for second dose of drug or placebo
* CVR < 1.4

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-04; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy M Crombleholme, MD, Principal Investigator — Children's Hospital of Cincinnati; Douglas Wilson, MD, Principal Investigator — Children's Hospital of Philadelphia; Hanmin Lee, MD, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - University of California, San Francisco Fetal Treatment Center, San Francisco, California
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Vu L, Tsao K, Lee H, Nobuhara K, Farmer D, Harrison M, Goldstein RB. Characteristics of congenital cystic adenomatoid malformations associated with nonimmune hydrops and outcome. J Pediatr Surg. 2007 Aug;42(8):1351-6. doi: 10.1016/j.jpedsurg.2007.03.039. PMID 17706495
- [Background] Schumacher A, Sidor J, Buhling KJ. [Continuous glucose monitoring using the glucose sensor CGMS in metabolically normal pregnant women during betamethasone therapy for fetal respiratory distress syndrome]. Z Geburtshilfe Neonatol. 2006 Oct;210(5):184-90. doi: 10.1055/s-2006-951743. German. PMID 17099841
- [Background] Peltoniemi OM, Kari MA, Tammela O, Lehtonen L, Marttila R, Halmesmaki E, Jouppila P, Hallman M; Repeat Antenatal Betamethasone Study Group. Randomized trial of a single repeat dose of prenatal betamethasone treatment in imminent preterm birth. Pediatrics. 2007 Feb;119(2):290-8. doi: 10.1542/peds.2006-1549. PMID 17272618
- [Background] Roberts D, Dalziel S. Antenatal corticosteroids for accelerating fetal lung maturation for women at risk of preterm birth. Cochrane Database Syst Rev. 2006 Jul 19;(3):CD004454. doi: 10.1002/14651858.CD004454.pub2. PMID 16856047
- [Background] Neilson JP. Antenatal corticosteroids for accelerating fetal lung maturation for women at risk of preterm birth. Obstet Gynecol. 2007 Jan;109(1):189-90. doi: 10.1097/01.aog.0000251610.51286.b1. No abstract available. PMID 17233108
- [Background] Tsao K, Hawgood S, Vu L, Hirose S, Sydorak R, Albanese CT, Farmer DL, Harrison MR, Lee H. Resolution of hydrops fetalis in congenital cystic adenomatoid malformation after prenatal steroid therapy. J Pediatr Surg. 2003 Mar;38(3):508-10. doi: 10.1053/jpsu.2003.50089. PMID 12632377
- [Background] Arca MJ, Teich S. Current controversies in perinatal care: fetal versus neonatal surgery. Clin Perinatol. 2004 Sep;31(3):629-48. doi: 10.1016/j.clp.2004.03.016. PMID 15325542
- [Background] Wilson RD, Baxter JK, Johnson MP, King M, Kasperski S, Crombleholme TM, Flake AW, Hedrick HL, Howell LJ, Adzick NS. Thoracoamniotic shunts: fetal treatment of pleural effusions and congenital cystic adenomatoid malformations. Fetal Diagn Ther. 2004 Sep-Oct;19(5):413-20. doi: 10.1159/000078994. PMID 15305098
- [Background] Knox EM, Kilby MD, Martin WL, Khan KS. In-utero pulmonary drainage in the management of primary hydrothorax and congenital cystic lung lesion: a systematic review. Ultrasound Obstet Gynecol. 2006 Oct;28(5):726-34. doi: 10.1002/uog.3812. PMID 17001747
- [Background] Davenport M, Warne SA, Cacciaguerra S, Patel S, Greenough A, Nicolaides K. Current outcome of antenally diagnosed cystic lung disease. J Pediatr Surg. 2004 Apr;39(4):549-56. doi: 10.1016/j.jpedsurg.2003.12.021. PMID 15065026
- [Background] Miller JA, Corteville JE, Langer JC. Congenital cystic adenomatoid malformation in the fetus: natural history and predictors of outcome. J Pediatr Surg. 1996 Jun;31(6):805-8. doi: 10.1016/s0022-3468(96)90138-4. PMID 8783108
- See also: Fetal Care Center of Cincinnati Children's Hospital — http://www.fetalcarecenter.org/
- See also: Fetal Treatment Center at the University of California, San Francisco — http://fetus.ucsfmedicalcenter.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only one participant was enrolled to the study before it was terminated; no participants were enrolled to the control arm
Period: Overall Study
Arm/Group | Active Study Group
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Only one participant was enrolled to the study before it was terminated; no participants were enrolled to the control arm
Arm/Group | Active Study Group
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Hydrops Fetalis
Time Frame: Delivery, up to approximately 20 weeks post-enrollment
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Active Study Group
Number analyzed (Participants) | 1
participants | 0

2. Secondary Outcome: Comparison of CCAM Size in Mid-trimester Fetuses (Study/Administration vs Control/Placebo)
Time Frame: Baseline, Delivery (up to approximately 20 weeks post-enrollment)
Population: Study was terminated without enrollment to control arm; therefore, no comparison was made
Arm/Group | Active Study Group
Number analyzed (Participants) | 0

3. Secondary Outcome: Survival at One-month Between Study and Control Groups.
Description: Status of neonate survival 30 days after delivery
Time Frame: 30 days after delivery (up to approximately 24 weeks post-enrollment)
Measure: Number; unit: participants
Arm/Group | Active Study Group
Number analyzed (Participants) | 1
participants | 1

ADVERSE EVENTS:
Time Frame: 30 days post-delivery (up to approximately 24 weeks)
Arm/Group | Active Study Group
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes